CLINICAL TRIAL: NCT02307318
Title: Heart and Hands Study II: A Retrospective Data Collection & Analysis Project
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HealthEast Care System (Other)
Collaborators: Chitogen, Inc. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H&H-002; Chit-002 (Other Grant/Funding Number: Chitogen, Inc)
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Thrombosis
Keywords: Radial Artery; Hemostasis; Angiography
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SoftSeal Hemostatic Pad (Other): This is a single arm study. All patients received the SoftSeal hemostatic pad for compression following elective or urgent coronary angiogram.
  Interventions: Device: SoftSeal Hemostatic Pad

INTERVENTIONS:
Device: SoftSeal Hemostatic Pad — Use of SoftSeal hemostatic device at a transradial access site with a 4 French system with with manual pressure by compression of the ulnar artery.

SUMMARY:
A recent pilot study conducted at HealthEast found use of manual pressure with the SoftSeal hemostatic pad for 15 minutes was successful in 9 out of 10 people fully anticoagluated using 4 French radial sheath. There was no evidence of radial artery occlusion in this small sample and bleeding was limited to grade 1. This evidence supports a larger retrospective study to confirm these results and define an alternative to the TR band use post radial artery access for cardiac catheterization.

Primary Objective Determine the incidence of arterial bleeding after real-world use of SoftSeal hemostatic device at a transradial access site with a 4 French system with with manual pressure by compression of the ulnar artery.

Secondary Objective Determine the incidence of thrombosis at the access site in all subjects as presence of thrombus in the radial artery by reverse barbeau test; the incidence of changes in circulation, movement and sensation (CMS) in the hand and wrist on the impacted hand; and the incidence of hematoma and ecchymosis, assessed just prior to discharge.

DETAILED DESCRIPTION:
This is a non-randomized, retrospective study to observe the usefulness of SoftSeal. Only patients with radial procedures will be used in this study.

Study Procedure For patients with a 4 French catheter, SoftSeal will be applied per physician instruction. Current protocol for use includes compression of ulnar artery on the same visit.

Any bleeding observed at the site after manual pressure hold with SoftSeal will constitute a failure to achieve hemostasis patient will be managed per standard of care (SOC).

Data Plan Following completion of clinical care we will extract data related to primary and secondary objectives. Data extraction will include documentation of CMS, reverse Barbeau and incidence of hematoma and ecchymosis. Any additional statistical analysis or manuscript writing will be done as part of a separate agreement to be met with the approval of both HaelaTheast Medical Research Institute and Chitogen.

Sample Size Calculation Since this is a real-world data analysis project with no control group, there is not a sample size calculation. We believe approximately 50 patients will be enough to provide an understanding of use instructions for the SoftSeal product.

ELIGIBILITY:
Inclusion Criteria:

* Transradial access site with a 4 French system ->18 years old

Exclusion Criteria:

* Current oral anti-coagulation therapy
* Prior participation in this study
* Positive standard-of-care pregnancy test
* Investigator discretionary exclusions
* Patient on dialysis
* GFR <30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Panetta, MD, Principal Investigator — HealthEast Care System
Locations (1):
- HealthEast Care System, Inc, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SoftSeal Hemostatic Pad: This is a single-arm study. All patients enrolled received the Softseal hemostatic pad for compression of the access site following elective or urgent coronary angiogram.
Period: Overall Study
Arm/Group | SoftSeal Hemostatic Pad
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SoftSeal Hemostatic Pad
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (8.7)
Gender [Count of Participants; unit: Participants]
  Female | 22
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Arterial Bleeding
Description: Number of patients who experience arterial bleeding after use of the Softseal hemostatic device and manual compression at the transradial access site as measured by observation.
Time Frame: Day1
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal Hemostatic Pad
Number analyzed (Participants) | 51
Participants | 1

2. Primary Outcome: Incidence of Thrombosis
Description: Number of patients who experience thrombosis (blood clot) at the access site as measured by ultrasound between 4 hours and 24 hours post-procedure.
Time Frame: 4 hours post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal Hemostatic Pad
Number analyzed (Participants) | 51
Participants | 0

3. Secondary Outcome: Changes in Circulation, Movement and Sensation
Description: Number of patients who experience changes in circulation, movement and sensation in the hand and wrist of the access site as measured by standard of care nursing assessments.
Time Frame: Day1
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal Hemostatic Pad
Number analyzed (Participants) | 51
Participants | 0

4. Secondary Outcome: Incidence of Hematoma and/or Ecchymosis
Description: Number of patients who experience hematoma (bruising) and/or ecchymosis (discoloration of the skin caused by bleeding underneath) at the access site as measured by observation just prior to discharge.
Time Frame: Day1
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal Hemostatic Pad
Number analyzed (Participants) | 51
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SoftSeal Hemostatic Pad
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No